CLINICAL TRIAL: NCT04845802
Title: Effects of Inspiratory Muscle Training on Diaphragm Thickness, Respiratory Muscle Strength and Balance in Dancers.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Hakan Aksu, PT, MSc Student in Exercise Physiology, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Iuhaksu01
Record Dates: First submitted 2021-04-12; First posted 2021-04-15 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Athletic Injuries
Keywords: Inspiratory Muscle Training; Diaphragm; Respiratory Muscle Strength; Balance; Dancer
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training Group (Experimental): Dancers in this group will perform inspiratory muscle training for 30 breaths, twice daily [morning: between 7:00 and 13:00 and evening: between 16:00 and 22:00], 7 days per week for 8 weeks, with a breathing frequency of 15 breaths per minute and a duty cycle of 0.5. One exercise session will be supervised in a clinic per week, other sessions will be performed at home in every week during the training.
  Interventions: Other: Inspiratory muscle training(high-IMT group)
- Sham Group (Sham Comparator): Dancers in this group will perform inspiratory muscle training for 30 breaths, twice daily [morning: between 7:00 and 13:00 and evening: between 16:00 and 22:00], 7 days per week for 8 weeks, with a breathing frequency of 15 breaths per minute and a duty cycle of 0.5. One exercise session will be supervised in a clinic per week, other sessions will be performed at home in every week during the training.
  Interventions: Other: Inspiratory muscle training(low-IMT group)

INTERVENTIONS:
Other: Inspiratory muscle training(high-IMT group) — A mechanical pressure threshold loading device (POWERbreathe, POWERbreathe International Ltd, UK) will be used for the training. Training intensity will set at 60% of the maximum inspiratory pressure.
  Other Names: [high-IMT group]
  Arms: Training Group
Other: Inspiratory muscle training(low-IMT group) — Dancers will be perform at a load setting of level 1 (corresponding to ~10% baseline MIP), using the same device as the training group.
  Other Names: [low-IMT group]
  Arms: Sham Group

SUMMARY:
Dance is a performing art form consisting of sports and art intertwined and complex dynamic choreographic figures were handled aesthetically and physically of narrative. Scientific studies are insufficient on dance and health and performance of dancers in the literature although dance is the most used type of art and sport in all societies and for all age groups. It is seen that the core stabilization (central forces) of the dancers is insufficient when the current studies were examined, this insufficient stabilization causes biomechanical changes in the trunk, and indirectly affects the lower extremities. Consequently, insufficient stabilization was shown to be caused impairment of force generation and injuries. In addition, lack of core stabilization of dancers may cause impairment in balance and postural control. Therefore, dancers need a good postural control with provided by an effective core stabilization training in order to exhibit a successful and healthy performance. It is shown that inspiratory muscle training (IMT) improves diaphragm strength and diaphragm thickness. Considering the relation between diaphragm muscle forming the upper (ceiling) part of the core area, and balance, IMT may also have an impact on postural control and balance alongside the standard clinical parameters such as respiratory muscle strength and diaphragm thickness in dancers. Thus, the aim of this study was to investigate the effects of inspiratory muscle training on diaphragm thickness, postural stability, balance, respiratory muscle strength in dancers.

ELIGIBILITY:
Inclusion Criteria:

* Dancer (for least two years)
* Stable clinical condition (no injury in last 2 months)

Exclusion Criteria:

* Documented diagnosis of vestibular, neurological or orthopedic disorders which may affect balance and mobility
* Having of chronic pulmonary disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Change of baseline postural stability test score in Biodex Balance System after 8 weeks | Eight weeks
  The Postural Stability Test evaluates static balance of participants. Postural Stability Test emphasizes a patient's ability to maintain center of balance. The patient's score on this test assesses deviations from center, thus a lower score is more desirable than a higher score.
Change of baseline athlete single leg stability score in Biodex Balance System after 8 weeks | Eight weeks
  The test protocol for the Athlete Single Leg Stability Testing allows clinicians to test athletes against data derived from studies using the Biodex Balance System. The stability level will challenge athletes and provide the data necessary to assess the athlete's single leg postural stability.
Change of baseline limits of stability test score in Biodex Balance System after 8 weeks | Eight weeks
  Limits of stability test evaluates dynamic balance of participants. Biodex balance system measures limits of stability for forward, backward, right and left side movements. It will calculate the maximum distance a person can lean without losing balance.
Change of baseline diaphragm thickness after 8 weeks | Eight weeks
  Two-dimensional B-mode ultrasound will be measure diaphragm thickness at the zone of apposition during inspiration or expiration using the intercostal approach. Diaphragm thickness will be measure as the vertical distance between the pleural and peritoneal layer at both Total Lung Capacity [TLC] and Functional Residual Capacity [FRC]. Measurements will be perform on the right hemidiaphragm with the volunteer in the supine position. All measurements will be perform 3 times and the average value for each calculate.
Change of baseline maximum inspiratory pressure after 8 weeks | Eight weeks
  Maximum inspiratory pressure (MIP) will be measure using a hand-held mouth pressure device. Three maximal manoeuvres will perform and the highest value record. Indirect measure of respiratory (inspiratory) muscle strength, expressed in cmH20.
Change of baseline maximum expiratory pressure after 8 weeks | Eight weeks
  Maximum expiratory pressure (MEP) will be measure using a hand-held mouth pressure device. Three maximal manoeuvres will perform and the highest value record. Indirect measure of respiratory (expiratory) muscle strength, expressed in cmH20.

SECONDARY OUTCOMES:
Change of baseline biering-sorenson test score after 8 weeks | Eight weeks
Change of baseline oswestry disability index after 8 weeks | Eight weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sensu Dincer, Dr., Principal Investigator — Istanbul University Faculty of Medicine Sports Medicine Department; Turker Sahinkaya, Lecturer, Principal Investigator — Istanbul University Faculty of Medicine Sports Medicine Department; Bulent Bayraktar, Prof. Dr., Study Director — Istanbul University Faculty of Medicine Sports Medicine Department

IPD SHARING:
Plan to Share IPD: Undecided
Patients may not want to share the data with anyone other than the researchers involved in the study.

REFERENCES:
- [Background] Janssens L, McConnell AK, Pijnenburg M, Claeys K, Goossens N, Lysens R, Troosters T, Brumagne S. Inspiratory muscle training affects proprioceptive use and low back pain. Med Sci Sports Exerc. 2015 Jan;47(1):12-9. doi: 10.1249/MSS.0000000000000385. PMID 24870567
- [Background] Ferraro FV, Gavin JP, Wainwright T, McConnell A. The effects of 8 weeks of inspiratory muscle training on the balance of healthy older adults: a randomized, double-blind, placebo-controlled study. Physiol Rep. 2019 May;7(9):e14076. doi: 10.14814/phy2.14076. PMID 31074198
- [Background] Watson T, Graning J, McPherson S, Carter E, Edwards J, Melcher I, Burgess T. DANCE, BALANCE AND CORE MUSCLE PERFORMANCE MEASURES ARE IMPROVED FOLLOWING A 9-WEEK CORE STABILIZATION TRAINING PROGRAM AMONG COMPETITIVE COLLEGIATE Dancers. Int J Sports Phys Ther. 2017 Feb;12(1):25-41. PMID 28217414